CLINICAL TRIAL: NCT02223988
Title: Occurrence of Ventilator Associated Pneumonia (VAP) in Italian ICU Using Cuffed Tracheostomy Tubes With Subglottic Secretion Drainage: a Prospective Observational Study.
Brief Title: Occurrence of Ventilator Associated Pneumonia in Italian ICU Using Cuffed Tracheostomy Tubes With Subglottic Secretion Drainage
Acronym: VICTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Marco Ranieri, MD, University of Turin, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CS/202
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Failure
Keywords: Patients; mechanical; ventilation; tracheostomy
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration

ARMS (1):
- subglottic secretion drainage (Experimental)
  Interventions: Procedure: subglottic secretion removal

INTERVENTIONS:
Procedure: subglottic secretion removal

SUMMARY:
Ventilator-associated pneumonia (VAP) is a serious complication and carries increased risks of morbidity and mortality for patients who require mechanical ventilation.

VAP is associated with the contamination and colonization of bacteria in the lower airway. These bacteria may be present in the lower airway by the aspiration of oropharyngeal secretions. Therefore limiting the amount of secretions that pass the glottis and enter the airway is paramount.

Patients who require prolonged mechanical ventilation may have a tracheostomy tube placed to manage breathing. These tubes may have a distal cuff which sits within the trachea. When the cuff is inflated, oropharyngeal secretions will pool above the cuff of the tracheostomy tube thereby limiting the amount of secretions entering the lower airway. These secretions may leak around the cuff and cause tracheobronchial colonization. It has been shown that removal of secretions that pool above the cuff via dorsal lumen suction leads to a decreased incidence of VAP.

The purpose of this study is to measure the effect of suction above the cuff tracheostomy tubes related to VAP incidence

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation for respiratory failure for at least 72 hours.
* A score of 35 to 65 on the Simplified Acute Physiology Score II (SAPS II).
* Does not have a pulmonary infection estimated by a Clinical Pulmonary Infection Score (CPIS).
* Age >= 18 years.
* have no exclusion criteria

Exclusion Criteria:

* A history of esophageal, tracheal or pulmonary cancer or an existing malignancy within the trachea at the tracheostomy site.
* Previous surgery at the tracheostomy site (e.g. thyroidectomy).
* Bleeding diathesis (e.g. due to anticoagulation therapy).
* Emergency surgical airway management.
* Morbid obesity and/or neck edema (skin to trachea distance may render tracheostomy tube too short).
* Pre-existing infection at the tracheostomy site.
* Uncertainty in identifying the anatomical landmarks.
* Patients with a do not resuscitate order.
* Immunosuppressed and/or immunodepressed patients (Immunodepression being defined by the following conditions: 1-Leukocytes < 1000/µl, 2-Neutrophils < 500/µl. 3-AIDS Long-term steroid treatment (daily dose > 0.5 mg/kg) for more than 30 days)
* Patients already enrolled in other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of VAP | at 28 days

SECONDARY OUTCOMES:
Mortality rate | at 28 days
  Mortality at 28-day (all-cause mortality) starting from enrollment (at tracheostomy time)
Duration of mechanical ventilation | 30 days
ICU length of stay | 30 days
Ventilator free days after tracheostomy | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pierpaolo Terragni, MD, Principal Investigator — Department of Anesthesia and Intensive Care Medicine, University of Turin, Italy
Locations (1):
- University of Turin - Department of Anesthesia and Intensive Care Medicine, Turin, Italy